CLINICAL TRIAL: NCT06126991
Title: Organ Protective Effect of Histamine H1 Receptor Antagonist In Patients With Severe Burns: A Clinical Study
Brief Title: Organ Protective Effect of Cetirizine In Patients With Severe Burns
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RuijinH_20230318
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-10

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Cetirizine; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Modified Sedation and Analgesia Regimen Group (Experimental): midazolam, fentanyl, cetirizine
  Interventions: Drug: Cetirizine; Drug: Midazolam and Fentanyl
- The Sedation and Analgesia Regimen Group (Active Comparator): midazolam, fentanyl
  Interventions: Drug: Midazolam and Fentanyl

INTERVENTIONS:
Drug: Cetirizine — Oral administration of cetirizine at 10mg once daily will be used.
  Arms: The Modified Sedation and Analgesia Regimen Group
Drug: Midazolam and Fentanyl — Midazolam 50mg + fentanyl 300ug micro pump push will be used with a starting dose of 5ml/hour, adjusted according to the patient's level of sedation. The patient's RASS score will be maintained between -1-0 and the drug will be suspended with a blood pressure below 90/60mmHg.

SUMMARY:
This prospective clinical trial aims to investigate the organ protective effects of cetirizine in patients with severe burns.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, parallel-controlled clinical trial. The global objective is to compare the organ protective effects of the sedation and analgesia regimen (midazolam, fentanyl) with the modified sedation and analgesia regimen (midazolam, fentanyl, cetirizine) in patients with severe burns (≥30% TBSA). Participants will receive the intervention from admission to 72 hours post-burn. Researchers will take the APACHE II scores on days 7 after admission as the main outcomes. Researchers will also take other supplementary examination results into account, including liver enzyme, myocardial enzyme, renal function, haemodynamic index, coagulation function, and pulmonary interstitial edema.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Commitment to comply with the procedures and cooperation during the course
* TBSA >30% and admitted within the first day after burns
* No severe compound injuries

Exclusion Criteria:

* History of allergy to drugs in the trial
* Postoperative complications that would interfere with the observation
* Mental illness and severe heart disease, hypertension
* Serious genetic diseases
* Incomplete clinical information (unclear diagnosis, incomplete medical history, incomplete medication records, etc.)
* Pregnancy/lactation
* Malignant tumors
* Organ insufficiency due to previous chronic diseases such as hypertension, diabetes mellitus or non-burning factors
* Serious adverse reactions
* Self-requested withdrawal

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
APACHE II on Day 7 | Day 7
  Observation of APACHE II scores of patients in each group 7 days after admission.
  The APACHE II (Acute Physiology And Chronic Health Evaluation II) is a severity-of-disease classification system. An integer score from 0 to 71 is computed based on several measurements. Higher scores correspond to more severe disease and a higher risk of death.

SECONDARY OUTCOMES:
Urinary Output | Day 7
  Observation of 24-hour urinary output (ml) 7 days after admission.
Blood L-lactate | Day 7
  Observation of Blood L-lactate level 7 days after admission.
Base Excess (BE) | Day 7
  Observation of base excess in blood 7 days after admission.
Oxygen Saturation | Day 7
  Observation of oxygen saturation in blood 7 days after admission.
Stroke Volume Variation | Day 7
  Observation of stroke volume variation (SVV) in PICCO or Uscom 7 days after admission.
Global End-Diastolic Volume | Day 7
  Observation of global end-diastolic volume (GEDV) in PICCO or Uscom 7 days after admission.
Central Venous Pressure | Day 7
  Observation of central venous pressure (CVP) in PICCO or Uscom 7 days after admission.
Stroke Volume | Day 7
  Observation of stroke volume 7 days after admission.
Cardiac Function Index | Day 7
  Observation of Cardiac Function Index (CFI) 7 days after admission.
Pulmonary interstitial edema | Day 7
  Observation of extravascular lung water index (ELWI) or chest x-ray 7 days after admission.
SOFA Score | Day 7
  Observation of SOFA score 7 days after admission.
  The SOFA score (Sequential Organ Failure Assessment Score) is a scoring system associated with the organ function or rate of function of patients. An integer score from 0 to 24 is computed based on 6 different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). Higher scores correspond to more severe organ function disorders or failures.
Body Temperature | Day 7
  Observation of body temperature 7 days after admission.
Heart Rate | Day 7
  Observation of heart rate 7 days after admission.
Respiratory Rate | Day 7
  Observation of respiratory rate 7 days after admission.
Leukocyte Count | Day 7
  Observation of leukocyte count in blood 7 days after admission.
Blood CRP | Day 7
  Observation of blood CRP (C-reactive protein) 7 days after admission.
Blood Calcitoninogen | Day 7
  Observation of blood calcitoninogen 7 days after admission.
Mechanical Ventilation Duration | Day 28
  Observation of mechanical ventilation duration during 28 days after admission.
Mortality | Day 28
  Observation of mortality during 28 days after admission.
Sepsis Rate | Day 28
  Observation of sepsis rate during 28 days after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Burn, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zhang M, Yang P, Yu T, Harmsen MC, Gao M, Liu D, Shi Y, Liu Y, Zhang X. Lytic cocktail: An effective method to alleviate severe burn induced hyper-metabolism through regulating white adipose tissue browning. Heliyon. 2022 Mar 17;8(3):e09128. doi: 10.1016/j.heliyon.2022.e09128. eCollection 2022 Mar. PMID 35846468
- [Result] Wang J, Lu C, Zhang J, Gao M, Liu D, Yang P, Yu T, Wang X, Zhang X, Liu Y. LYTIC COCKTAIL ATTENUATES CATECHOLAMINE SURGE AFTER SEVERE BURNS BY BLOCKING HISTAMINE H1 RECEPTOR/PKA/CREB/TYROSINE HYDROXYLASE SIGNALING IN CHROMAFFIN CELLS. Shock. 2022 Aug 1;58(2):158-168. doi: 10.1097/SHK.0000000000001963. Epub 2022 Jul 24. PMID 35953455
- [Result] Wang J, Lu C, Liu X, Zhang G, Zhang J, Gao M, Liu D, Zhang X, Liu Y. Histamine H1 receptor antagonist attenuates catecholamine surge and organ injury after severe burns. Front Endocrinol (Lausanne). 2023 Feb 9;14:1068925. doi: 10.3389/fendo.2023.1068925. eCollection 2023. PMID 36843581